CLINICAL TRIAL: NCT00482001
Title: The Impact of Cholinesterase Inhibitors on Driving Ability in Healthy Older Adults: A Pilot Study
Brief Title: Impact of Cholinesterase Inhibitors on Driving Ability in Healthy Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 458970
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Mental Health; Geriatrics
Keywords: Donepezil; Driving; Cholinesterase Inhibitors; Geriatric Psychiatry; Psychopharmacology; Aricept
MeSH Terms: conditions — Psychological Well-Being | interventions — Donepezil; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- donepezil (Experimental): donepezil, capsule, 5mg daily once daily for 14 days
  Interventions: Drug: donepezil
- placebo (Placebo Comparator): placebo (cornstarch), capsule, once daily for 14 days
  Interventions: Drug: Placebo (cornstarch)

INTERVENTIONS:
Drug: donepezil
  Other Names: Aricept
  Arms: donepezil
Drug: Placebo (cornstarch)
  Arms: placebo

SUMMARY:
The goal of the study is to assess the role of cholinesterase inhibitors in affecting the driving ability of cognitively intact seniors using driving simulators. We hypothesize that the use of a cholinesterase inhibitor for two weeks will be associated with improvement in safe driving behavior on a simulated driving task.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia, and while it is known that AD poses substantial risks of motor vehicle collisions, many people in the earliest stages of AD continue to drive. Memory problems themselves are poor predictors of who is actually unsafe on the road, and various medications that are used to treat people with AD may impact on their driving abilities. Donepezil is a drug used to treat the memory problems associated with AD. While previous studies have shown that it slows the decline of activities of daily living (eg. shopping, banking, dressing) and may improve the ability of younger pilots to perform on computerized flight simulators, no studies have examined the impact of donepezil on driving abilities in older adults.

The present investigation is a pilot study aiming to determine if donepezil helps healthy older drivers perform on driving simulators. Two Canadian academic centers have different driving simulators - one in Toronto and one in Thunder Bay. At each of these centers, ten healthy men aged 65 to 75 will be randomly assigned to receive either donepezil 5mg/day or identical placebo for two weeks.

Using the driving simulator, we will assess various aspects of driving ability. These measures of driving performance will be compared between those who received the drug and those who received the placebo.

ELIGIBILITY:
Inclusion Criteria:

* valid Ontario driver's license
* active driver (greater than or equal to three times per week)
* written, informed consent
* lives in Toronto/Thunder Bay
* healthy
* Male between 65-75 years old

Exclusion Criteria:

* cognitive impairment
* psychiatric history
* sleep disorder history
* substance abuse
* neurological history
* medical illness
* ophthalmological disease
* psychoactive medications
* contra-indications to Donepezil
* experience car/motion sickness

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rapoport, MD, FRCPC, Principal Investigator — University of Toronto; Michel Bedard, PhD, Study Chair — Lakehead University; Nathan Herrmann, MD, FRCPC, Study Chair — University of Toronto; Krista Lanctot, PhD, Study Chair — University of Toronto
Locations (2):
- Canada (2):
  - Lakehead University, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: donepezil: donepezil 5mg, once daily for 2 weeks
- Placebo: Placebo (cornstarch): 1 capsule daily for 2 weeks
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.6) | 70.8 (4.7) | 71.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 10 | 20
number of driving days/week [Mean (Standard Deviation); unit: days] | 6.55 (1.0) | 5.80 (1.6) | 6.18 (1.35)
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE), range 0-30, with higher scores indicating better mental state/ cognitive performance
  units on a scale | 29.30 (1.1) | 29.50 (0.7) | 29.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Test (PVT)
Description: A measure of reaction time in milliseconds, using a handheld unit, in which participants respond to a visual simulus
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
milliseconds | 302.62 (53.0) | 277.13 (23.9)

2. Primary Outcome: Attention Network Test (ANT)
Description: A measure of reaction time in milliseconds, based on the speed with which participants press a key in response to a visual stimulus
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Donepezil: donepezil, capsule, 5mg daily once daily for 14 days
  donepezil
- Placebo: placebo (cornstarch), capsule, once daily for 14 days
  Placebo (cornstarch)
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
milliseconds | 672.37 (70.9) | 637.58 (68.7)

3. Primary Outcome: Speed Deviation
Description: A measure of deviation from posted speed limit, measured in km/h
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: kilometers / hour
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
kilometers / hour | -1.09 (6.6) | -2.41 (4.8)

4. Primary Outcome: Deviation From Road Position
Description: A measure of deviation from central road position, measured in cm
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
centimeters | 27.54 (1.1) | 26.06 (1.7)

5. Primary Outcome: Reaction Time to Wind Gusts
Description: Reaction time to wind gusts, measured in seconds
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
seconds | 1.69 (0.5) | 1.18 (0.3)

6. Primary Outcome: Percentage of Time in Safe Zone
Description: Time spent in safe zone (within 10km/h of speed limit and within 0.838m of centre of driving lane), measured as %
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 60.95 (21.4) | 74.79 (17.6)

7. Primary Outcome: Collisions
Description: Number of collisions (on driving simulator)
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: collisions
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
collisions | 0.40 (0.7) | 0.30 (0.5)

ADVERSE EVENTS:
Time Frame: Day 8
Groups:
- Donepezil: donepezil 5mg, one capsule daily for 14 days
- Placebo: Placebo (cornstarch), 1 capsule daily for 14 days
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=11) | Placebo (N=11)
anorexia (General disorders) | 0 (0) | 1 (1)
nausea / diarrhea (General disorders) | 1 (1) | 0 (0)
fatigue / somnolence (General disorders) | 2 (2) | 2 (2)
headaches / abnormal dreams (General disorders) | 2 (2) | 1 (1)
insomnia (General disorders) | 1 (1) | 0 (0)
frequent urination (General disorders) | 5 (5) | 0 (0)
thirst (General disorders) | 0 (0) | 1 (1)
rash (General disorders) | 0 (0) | 1 (1)
dry mouth (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No